CLINICAL TRIAL: NCT06595407
Title: Loss of Y Chromosome in Aortic Stenosis
Status: Recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jonathan Lindner, MD, Professor of Medicine, University of Virginia
Other Study IDs: 301597
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Aortic Stenosis
Keywords: Aortic stenosis; Y-chromosome; Transforming growth factor-beta; Echocardiography
MeSH Terms: conditions — Aortic Valve Stenosis; Camurati-Engelmann Syndrome | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples containing leukocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Males with aortic stenosis: Males with mild or greater aortic stenosis (aortic valve area <1.5 cm2) due to calcific non-congenital aortic stenosis.
  Interventions: Diagnostic Test: Blood analysis for loss-of-Y chromosome
- Control males without aortic stenosis: Males without any diagnosis for aortic stenosis (matched for aortic stenosis group).
  Interventions: Diagnostic Test: Blood analysis for loss-of-Y chromosome

INTERVENTIONS:
Diagnostic Test: Blood analysis for loss-of-Y chromosome — Analysis for the percentage of circulating leukocytes with loss-of-y chromosome

SUMMARY:
The most common heart valve disease in humans is aortic stenosis which is a critical narrowing of the valve through which the heart has to pump blood to the rest of the body. This condition occurs in 2-3% of adults over 65 years of age and when it progresses to a severe stage leads to heart failure and need for valve replacement procedures (including surgery and catheter-based replacement). Aortic stenosis has a strong male predominance. The purpose of this study is to evaluate whether loss of Y-chromosome from circulating blood cells in males, which has been associated with TGF-beta-related fibrosis of other organs, is associated with the development of aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Aortic stenosis (valve area <1.5cm2)

Exclusion Criteria:

* Bicuspid aortic valve
* History of radiation to chest
* Inflammatory (autoimmune, rheumatologic) disease associated with aortic stenosis
* Active cancer

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males with calcific, non-congenital aortic stenosis and age-matched males without aortic stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Loss of Y chromosome | 1 day
  This is a cross-sectional case-control study where the outcome measure is the percentage of circulating cells that have loss-of-Y chromosome

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
All data generated during the course of this research will be made available in accordance with the Final NIH Statement of Sharing Research Data, Notice: NOT-OD-03-032. Data will be shared on the common data elements (CDE) system from the NIH CDE Repository.
Supporting Information: Study Protocol, ICF
Access Criteria: Open access